CLINICAL TRIAL: NCT07132788
Title: Understanding the Effects of Pulmonary Arterial Hypertension on Lean Muscle Mass
Acronym: MUSCLE UP-PH
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 856202; R01HL173533 (NIH)
Record Dates: First submitted 2025-07-01; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; body composition
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Blood Specimen Collection; Walk Test; Absorptiometry, Photon; Echocardiography; Caves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood draw — Research blood draw
Diagnostic Test: Short Performance Physical Battery — test of physical performance, which involves measuring movement from sitting to standing, walking speed, and balance
Diagnostic Test: Grip strength test — Measures grip strength
Diagnostic Test: Six minute walk test — Measures distance walked in 6 minutes
Radiation: Chest CT scan — X-ray and computer technology takes detailed pictures of the organs and structures inside your chest
Radiation: Dual-Energy X-ray Absorptiometry Scan — Uses X-ray technology to measure the mineral density of your bones, and provides a ratio of fat tissue to lean mass (muscle) and bone
  Other Names: DXA Scan; DEXA Scan
Behavioral: Activity monitoring — A device worn on your non-dominant wrist which measures motion/ movement/ activity
Behavioral: 24 hour diet recall — A research dietitian will contact you and ask you to provide details of what you ate over the previous 24 hours
Diagnostic Test: Echocardiogram — Ultrasound technology to create moving images of your heart, valves, and chambers
  Other Names: Echo; Cardiac Ultrasound
Behavioral: Quality of Life Questionnaire (emPHasis 10) — The emPHasis-10 is a pulmonary hypertension-specific questionnaire which is scored from 0-50 (with higher scores indicating worse quality of life.)
  Other Names: emPHasis 10
Behavioral: International Physical Activity Questionnaire Short Form (IPAQ-SF) — The IPAQ-SF is a small set of questions to obtain comparable estimates of physical activity.
  Other Names: IPAQ-SF

SUMMARY:
Patients with pulmonary arterial hypertension (PAH) are at increased risk of muscle loss and decreased physical activity. This study will aim to (1) understand the way in which muscle loss occurs in PAH, particularly the role of fat surrounding the heart, and (2) look at the impact muscle loss has on quality of life, daily physical activity, and hospitalizations in patients with PAH. The findings from this study could help identify potentially treatable factors that may improve the overall quality of life and physical functioning of patients with PAH.

Subjects will be asked to attend a baseline visit where the following will be performed:

* Measure your vital signs
* Undergo a research blood draw, less than 4 tablespoons
* Provide a urine pregnancy test (if applicable)
* Review demographics, personal history, and medical history
* Review current PAH medications
* Complete questionnaires on how your PAH affects you
* Complete a test of physical performance
* Complete a grip strength test
* Undergo an echocardiogram (Echo)
* Complete a six-minute walk test
* Undergo a Chest CT Scan
* Undergo a scan of your body composition (DXA scan)
* Obtain a weight and body composition measurement on the InBody Scale Subjects will also complete activity moniotring, two 24-hour diet recalls, and participate in remote follow-up visits every 6 months

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study mandated procedure.
* Diagnosis of PAH belonging to one of the following subgroups of Group 1 PH according to the updated clinical classification [Humbert 2022]

  * Idiopathic (IPAH)
  * Heritable (HPAH)
  * Drugs or toxins induced
  * Associated (APAH) with one of the following:

    * Connective tissue disease;
    * Human immunodeficiency virus (HIV) infection;
    * Congenital heart disease; or
    * Portopulmonary hypertension
* Diagnosis of PAH within 6 months of enrollment or diagnosis of PAH and on stable therapy for 3 months prior to enrollment
* Documented hemodynamic diagnosis of PAH by right heart catheterization (RHC), prior to enrollment showing:

  * mPAP > 20 mmHg; and
  * PAWP or LVEDP ≤ 15 mmHg
  * PVR > 2 Wood units

Exclusion Criteria:

* Prior to enrollment, evidence of moderately severe obstructive ventilator defect with:

  * FEV1/FVC ≤ 5th percentile; and
  * FEV1 z-score < 2.5
* Prior to enrollment, evidence of severe restrictive defect with

  * TLC < 5th percentile
  * FEV1 z-score < 4
* Prior to enrollment, hospitalization (within 1 week) for decompensated right heart failure
* More than moderate aortic or mitral valve disease
* LVEF < 40% within 1 year of screening
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include Pulmonary Hypertension patients from the University of Pennsylvania and Rhode Island Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Intake of food and nutrients | One time at Baseline
  Adequacy of micronutrient and protein intake are derived from the two 24 hour diets recalls.
Epicardial adipose tissue (EAT) volume | One time at Baseline
  Derived from chest CT
Metabolomics | One time at Baseline
  Circulating proteins will be measured in plasma samples using the Olink Proteomics (Waltham, MA). In this assay, Olink uses a proprietary proximity extension assay technology to combine a detection step involving oligonucleotide-labeled antibodies with a proximity-dependent DNA polymerization step and a real-time quantitative PCR amplification step to measure relative levels of multiple biomarkers simultaneously. Two different panels will be used: Olink Explore 384 Cardiometabolic and Olink Explore 384 Inflammation.
Right ventricular (RV) function | One time at Baseline
  Determined from 2D echocardiography
Adiponectin | One time at Baseline
  Measured using a solid phase sandwich ELISA (R&D Systems, Inc., Minneapolis, MN) with a minimum detectable dose of 0.246 ng/mL and intra-assay variations (CV) 2.5%-4.7%.
Low lean mass | One time at Baseline
  Using the data from the dual-energy X-ray absorptiometry, we will generate fat mass index-adjusted appendicular lean mass index (ALMIFMI) Z-Scores derived from age, sex, and race/ethnicity specific models.16 Low lean mass will be defined as ALMIFMI ZScore less than or equal to -1.
Accelerometry measures | One time at Baseline
  Step counts and activity intensity (sedentary time, time spent doing light, moderate, and vigorous activity) will be derived.
Health-Related Quality of Life (HRQOL) | One time at Baseline
  The emPHasis-10 is a questionnaire used to assess the impact of pulmonary hypertension (PH) on a person's life. It consists of 10 items, each scored on a scale of 0 to 5, resulting in a total score ranging from 0 to 50. Higher scores indicate a greater symptom burden and poorer quality of life.

SECONDARY OUTCOMES:
Chest Computed Tomographic (CT) scan | One time at Baseline
  The primary variables of interest will be total thoracic muscle volume measured on non-contrast chest CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Al-Naamani, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Hospital, Philadelphia, Pennsylvania, United States